CLINICAL TRIAL: NCT06201429
Title: A Multi-center, Early Feasibility Study of Using the Mechanical Tissue Resuscitation™ (MTR™) Therapy System for Removal of Excess Fluid in Subjects Who Have Had a Portion of Their Skull Removed to Expose the Dura/Brain and Require Drainage for Fluid Removal.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Renovo Concepts, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2023-01
Record Dates: First submitted 2023-12-30; First posted 2024-01-11 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Clinical Need for Craniotomy or Craniectomy
Keywords: craniotomy; craniectomy

STUDY DESIGN:
Intervention Model Description: Single arm early feasibility study. The study will comprise of patients who will receive MTR™ therapy to remove fluid from the surgical site in patients that have undergone a craniotomy/craniectomy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Mechanical Tissue Resuscitation (MTR™) (Experimental)
  Interventions: Device: Mechanical Tissue Resuscitation (MTR™)

INTERVENTIONS:
Device: Mechanical Tissue Resuscitation (MTR™) — Mechanical Tissue Resuscitation (MTR™) to externally drain excess fluid volume from the site of surgery in patients who have undergone a surgical procedure (craniotomy/craniectomy) for which a portion of the skull has been removed resulting in exposure of the dura/brain and require drainage of fluid.

SUMMARY:
A multi-center, early feasibility study of using the Mechanical Tissue Resuscitation™ (MTR™) therapy system for removal of excess fluid in subjects who have had a portion of their skull removed to expose the dura/brain and require drainage for fluid removal.

DETAILED DESCRIPTION:
Mechanical Tissue Resuscitation (MTR™) is intended for short-term (up to 7 days) use to externally drain excess fluid volume from the site of surgery in patients who have undergone a surgical procedure (craniotomy/craniectomy) for which a portion of the skull has been removed resulting in exposure of the dura/brain and require drainage of fluid.

This is a single arm early feasibility study. The study will comprise of patients who will receive MTR™ therapy to remove fluid from the surgical site in patients that have undergone a craniotomy/craniectomy.

The patient population will include male and female patients ages 22-65 who have undergone a surgical procedure to remove a portion of the skull to expose the dura/brain (craniotomy or craniectomy) in which the dura is intact or has been closed (repaired), and who, as an integral part of their care would require placement of a Jackson Pratt drain.

Patients will be treated with MTR™ for up to seven (7) days, with a follow up evaluation approximately one month post treatment.

Patients who have suffered a traumatic brain injury (TBI) and require such a surgical procedure are not to be included in the patient population for this early feasibility study.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is willing and able to provide written informed consent.
2. The patient's age is ≥ 22 and ≤ 65 years.
3. The patient has a clinical need for a craniotomy/craniectomy and for which, as an integral part of their care, a Jackson Pratt (JP) drain would be placed at the surgical site.
4. The surgical case is classified as 'clean'.

Exclusion Criteria:

1. Patient has suffered a traumatic brain injury.
2. Patient is pregnant or lactating.
3. Patient's BMI = (Weight (lb) x 703)/(〖Height〗^2 (inches)) > 45; BMI may also be calculated at http://nhlbi.nih.gov/health/educational/lose_wt/BMI/bmicalc.htm
4. Patient is participating in another clinical investigation .
5. Patient's anticipated survival is < 48 hours.
6. Patient is incarcerated at time of hospital admission.
7. Patient has a coincidental infection.
8. Patient has thrombocytopenia (platelet count < 150,000/µL).
9. Patient has an International Normalized Ratio (INR) > 1.5.
10. Patient is an active opioid abuser.
11. Patient is an active alcohol abuser.
12. There is active bleeding at the site of surgery.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2024-01-15 (Estimated); Primary Completion 2024-04-15 (Estimated); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
Safety and effectiveness of MTR™ | 30 days
  The primary endpoint is to evaluate MTR™ as safe and effective for the removal of fluids in those patients who have undergone a craniotomy/craniectomy, and to assess the frequency of device and procedure related adverse events.

SECONDARY OUTCOMES:
MTR™ Success | 30 days
  MTR™ Success will be defined as:
  1. Placement: ability to establish and maintain pressure with adequate manifold sizing.
  2. Maintenance: lack of air leaks and evidence of fluid removal.
  3. Removal: ability to remove without tissue damage or excessive bleeding.
AEs/SAEs Frequency | 30 days
  Frequency of all adverse events experienced from the time of enrollment through study exit. Events will be categorized as adverse events (AEs) or serious adverse events (SAEs) and measured by site data entry review.
Ability to remove fluid | 7 days
  Ability to remove fluid, measured volume of fluid and rate of removal.
Operator ease survey | 1 day (during day of surgery)
  Operator survey measured by completion of the following 3 questions on the case report form for:
  1. ease of manifold placement,
  2. ease of exit tubing placement,
  3. ease of establishment of a vacuum seal.
  Answered with a five category Likert scale ranging from Extremely Easy to Extremely Difficult.
Health care professional (HCP) ease survey | 1 day (during day of surgery)
  HCP survey regarding ease of system use/maintenance during treatment period.
  Answered with a four category Likert scale ranging from Poor to Excellent for each specific category below:
  1. MTR Manifold (silicone foam) Sheet Placement
  2. Dome and Tubing Assembly Placement
  3. Use of Sub-Atmospheric Pressure Pump (SaPP™)
  4. Vacuum - Site closure
  5. Fluid Removal
Data Integrity | 30 days
  Data integrity measured by the frequency of each type of missing data query seen during the course of the subject's treatment, and frequency of any other protocol deviation recorded during the study.

IPD SHARING:
Plan to Share IPD: No